CLINICAL TRIAL: NCT02932267
Title: Subject Reported Outcomes With Use of Adapalene 0.3% - Benzoyl Peroxide 2.5% in Moderate to Severe Acne in Dark Skin Phototype Subjects
Brief Title: Subject Reported Outcomes With Use of Adapalene 0.3% - Benzoyl Peroxide (BPO) 2.5% in Dark Skin Acne
Acronym: EDeN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.03.SPR.110232
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2019-12

CONDITIONS: Acne Vulgaris
Keywords: Acne; Dark skin
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Gels; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adapalene / BPO gel (Experimental): Adapalene 0.3% / BPO 2.5% gel, once daily in the evening
  Interventions: Drug: Adapalene 0.3% / BPO 2.5% gel

INTERVENTIONS:
Drug: Adapalene 0.3% / BPO 2.5% gel — Epiduo Forte / Tactupump gel to be applied once a daily at bed time on entire face during 16 weeks
  Other Names: Epiduo Forte / Tactupump gel

SUMMARY:
This is a multicenter open-label, prospective study in subjects with dark skin from one of the 3 ethnic/race backgrounds: Asian, Latin American and Black/African-American and with moderate to severe acne vulgaris on the face.

All eligible subjects will receive Adapalene 0.3% - BPO 2.5% gel (Epiduo Forte/TactuPump Forte) once daily on whole face.

The purpose of this trial is to evaluate subject reported outcomes with the combination of Adapalene 0.3% - BPO 2.5%, Epiduo Forte / TactuPump Forte gel, after 16 weeks of treatment of moderate to severe acne in dark skin phototypes (IV to VI).

ELIGIBILITY:
Inclusion Criteria:

* Subject with clinical diagnosis of moderate to severe facial acne vulgaris, defined by:

  1. Investigator's Global Assessment (IGA) score of 3 (Moderate) OR 4 (Severe ); and
  2. A minimum of 25-100 inflammatory lesions (papules and pustules); and
  3. A minimum of 30-150 non-inflammatory lesions (open and closed comedones) in total (excluding the nose); and
  4. No more than two acne nodules (≥ 1 cm),
* Subject with skin phototype IV to VI on Fitzpatrick skin phototype scale,
* Subjects from one of the 3 ethnic/race backgrounds: Asian, Latin American and Black/African-American,

Exclusion Criteria:

* Subject with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), nodulo cystic acne, acne requiring systemic treatment,
* Subject with history of lupus, atopic dermatitis, perioral dermatitis, dermatomyositis, rosacea
* Female subject who is pregnant, lactating or planning a pregnancy during the trial,
* Subjects having received at least one of the following topical treatments on the treated area: Corticosteroids, antibiotics, benzoyl peroxide, azelaic acid, dapsone, hydroxyacids, Zinc containing treatments, antiseptics, other anti-inflammatory products or other acne treatments (2 weeks); Retinoids (4 weeks); Cosmetic/aesthetic procedures on the face (1 week); Wax epilation (2 weeks); Photodynamic therapy (6 weeks); Laser therapy, microdermabrasion, deep chemical peel, plastic surgery for acne (3 months).
* Subjects having received at least one of the following systemic treatments: Corticosteroids, tetracyclines, other antibiotics (except penicillin) (1 month); Oral retinoids/isotretinoin/ anti-androgens / Cyproterone acetate / Chlormadinone acetate (6 months); Spironolactone/ Drospirenone (3 months); Immunomodulators (3 months) and Oral contraceptives/ oral dapsone for acne(1 month).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Dermresearch, Austin, Texas, United States
- CIDP, Phoenix, Mauritius
- CIDP, Singapore, Singapore

REFERENCES:
- [Derived] DuBois J, Ong GCW, Petkar G, Almeida LMC, Chavda R, Kerrouche N, Alexis AF. Patient-Reported Outcomes in Acne Patients With Skin of Color Using Adapalene 0.3%-Benzoyl Peroxide 2.5%: A Prospective Real-World Study. J Drugs Dermatol. 2019 Jun 1;18(5):514. PMID 31251543

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Wash-out period for topical treatment or procedures of 1 week to 3 months and for systemic treatment for 1 month to 3 months, depending on treatment
Period: Overall Study
Arm/Group | Adapalene / BPO Gel
Started | 50
Completed | 42
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 4
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Arm/Group | Adapalene / BPO Gel
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20
  Latin American | 13
  Black/African-American | 17
Region of Enrollment [Number; unit: participants]
  Singapore | 16
  United States | 18
  Mauritius | 16
Skin phototype [Count of Participants; unit: Participants] — Fitzpatrick skin phototype is a system used to describe a person's skin type. It ranges from skin phototype I to VI. Where, skin phototype I = pale white skin, always burns easily, never tans; skin phototype II = fair skin, always burns easily, tans minimally and with difficulty; skin phototype III = darker white skin, burns minimally, tans gradually and uniformly; skin phototype IV = light brown skin, burns minimally, always tans well; skin phototype V = brown skin, rarely burns, tans profusely; skin phototype VI = dark brown or black skin, never burns, tans profusely.
  Participants
    Phototype IV | 37
    Phototype V | 11
    Phototype VI | 2

OUTCOME MEASURES:

1. Primary Outcome: Subject 's Overall Satisfaction With Study Treatment Via a Satisfaction Questionnaire
Description: % of subjects satisfied to very satisfied with study treatment at week 12
Time Frame: At week 12
Population: Intent-to-treat (ITT) population. Here 'N' (number analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene / BPO Gel
Number analyzed (Participants) | 47
Participants | 36

ADVERSE EVENTS:
Time Frame: Up to 16 Weeks
Arm/Group | Adapalene / BPO Gel
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 9/50
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene / BPO Gel (N=50)
Pyrexia (General disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (4)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Version for USA (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT02932267/Prot_SAP_000.pdf